CLINICAL TRIAL: NCT04115800
Title: Subconjunctival Treatment of Liposomal Sirolimus as a Treatment for Dry Eye Disease
Brief Title: Liposomal Sirolimus in Dry Eye Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI-2019/04/01
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Dry Eye
Keywords: Sirolimus; Liposomal; Subconjunctival
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Sirolimus (Experimental): Subconjunctival injections of liposomal sirolimus in patients with conventional treatment with moderate and severe dry deye disease
  Interventions: Drug: Liposomal Sirolimus
- Liposomal (Placebo Comparator): Subconjunctival liposomal injections in patients with conventional treatments and moderate and severe dry eye disease
  Interventions: Drug: Liposomal Sirolimus

INTERVENTIONS:
Drug: Liposomal Sirolimus — Subconjunctival injections of liposomal sirolimus in patients with conventional treatment with moderate and severe dry deye disease

SUMMARY:
Dry eye disease is a very frequent pathology that importantly affects the quality of life of patients; in spite of the common use of eye lubricants to ameliorate symptoms, there is still a large number of patients who do not present improvement of the disease or they worsen. Although its etiology is varied, the imbalance of the immune system plays a substantial role in the development of dry eye disease. Rapamycin or sirolimus is an anti-inflammatory and immunomodulatory drug that has an enormous potential in ocular surface pathologies such as dry eye disease. The aim of the present study is to determine the effectiveness and security of subconjunctival application of a new formulated drug of liposomal sirolimus in patients with moderate and severe dry eye disease. This is a randomized placebo-controlled double blind clinical trial. Patients presenting data of moderate or severe dry eye disease will be randomized into two groups. One group will receive additional to the conventional treatment, subconjunctival injections of liposomal sirolimus; meanwhile the other group will receive subconjunctival placebo injections. After intervention the effectiveness and the security of the liposomal sirolimus will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate or severe Dry Eye
* Subjects with OSDI score > 22
* Subjects with Van Bijsterveld staining score >4
* Subjects that accept to participate in the study

Exclusion Criteria:

* Subjects with refraction surgery antecedents
* Subjects with ophthalmic surgery six months previous to the study
* Subjects with Lagophthalmos
* Subjects with facial paralysis antecedents
* Subjects with herpetic keratitis
* Subjects using isotretinoin
* Pregnant subjects
* Subjects in lactating period
* Subjects with allergy or intolerant to the drug
* Subjects with hepatic disorders
* Subjects with abnormal thoracic X rays

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Six weeks after intervention
  The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal patients and patients with dry eye disease. The OSDI is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and sever) and effect on vision -related function.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided